CLINICAL TRIAL: NCT06255977
Title: A Multicenter, Randomized, Blind, Placebo-controlled, Dose-finding Phase II Trial Evaluating the Safety and Efficacy of the Neuroprotective Peptide CN-105 in Patients With Acute Supratentorial Intracerebral Hemorrhage (CN-CATCH)
Brief Title: A Study Evaluating the Safety and Efficacy of Neuroprotective Peptide CN-105 Peptide in Patients With Acute Supratentorial Intracerebral Hemorrhage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: SDM Bio Service Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-CBT-2019040-2F
Record Dates: First submitted 2023-12-24; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — apolipoprotein E mimetic peptide CN-105

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Control: placebo (Placebo Comparator): Intravenous infusion with placebo（same volume of saline） every 6 hours, up to a maximum of 13 doses within 72 hours.Each dose of placebo（same volume of saline） will be administered as a slow IV bolus over 30 minutes.
  Interventions: Drug: CN-105
- Experimental: CN-105 peptide for injection 0.1 mg/kg (Experimental): Intravenous infusion with 0.1 mg/kg CN-105 peptide for injection every 6 hours, up to a maximum of 13 doses within 72 hours.Each dose of CN-105 will be administered as a slow IV bolus over 30 minutes.
  Interventions: Drug: CN-105
- Experimental:CN-105 peptide for injection 0.3 mg/kg (Experimental): Intravenous infusion with 0.3 mg/kg CN-105 peptide for injection every 6 hours, up to a maximum of 13 doses within 72 hours.Each dose of CN-105 will be administered as a slow IV bolus over 30 minutes.
  Interventions: Drug: CN-105
- Experimental: CN-105 peptide for injection 1.0 mg/kg (Experimental): Intravenous infusion with 1.0 mg/kg CN-105 peptide for injection every 6 hours, up to a maximum of 13 doses within 72 hours.Each dose of CN-105 will be administered as a slow IV bolus over 30 minutes.
  Interventions: Drug: CN-105

INTERVENTIONS:
Drug: CN-105 — Injection every 6 hours, up to a maximum of 13 doses within 72 hours.Each dose of CN-105 will be administered as a slow IV bolus over 30 minutes.
  Other Names: CN-105peptide

SUMMARY:
Intracerebral hemorrhage (ICH) is a devastating form of cerebrovascular disease for which there are no approved therapeutics that improve outcomes. Apolipoprotein E (apoE) has emerged as a promising therapeutic target given its isoform-specific neuroprotective properties and ability to modulate neuroinflammatory responses. We developed a 5-amino acid peptide, CN-105, that mimics the polar face of the apoE helical domain involved in receptor interactions, readily crosses the blood-brain barrier, and improves outcomes in well-established preclinical ICH models. In the current study, aim to assess the safety and the efficacy of CN-105 after administration for three consecutive days in participants with acute supratentorial ICH at three different dosages.

DETAILED DESCRIPTION:
Inclusion Patients with spontaneous acute supratentorial intracerebral hemorrhage confirmed by CT，age 30 to 80 years，Intravenous infusion with CN-105 peptide for injection every 6 hours, up to a maximum of 13 doses within 72 hours。

Blood samples for protein markers will be collected and detected at screening, 48 h(D3), and 120 h(D6) after the first dose:

The sample size is 240.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, age 30 to 80 years, inclusive;
2. Has a confirmed diagnosis of spontaneous supratentorial ICH by CT;
3. Able to receive first dose of study drug ≤ 12 hours after onset of ICH symptoms, such as alteration in level of consciousness, severe headache, nausea, vomiting, seizure, and/or focal neurological deficits, or last-known well time;
4. Has a GCS score ≥ 8 at enrollment;
5. Has an NIHSS score ≥ 6
6. Has Systolic BP (SBP) < 200 mmHg
7. Has given written informed consent to participate in the study in accordance with required regulations; if a participant is not capable of providing informed consent, written consent must be obtained from the participant's legally authorized representative (LAR).

Exclusion Criteria:

1. Is pregnant or lactating;
2. Has a temperature greater than 38.5℃ at Screening;
3. The amount of intracerebral hemorrhage< 5 mL（ coniglobus formula）
4. ICH known to result from trauma;
5. Primary intraventricular hemorrhage；
6. Radiographic evidence of underlying brain tumor;
7. Patients with a history of malignant tumor (non-melanoma in situ skin cancer that has achieved complete remission after treatment and has not relapsed in the past 5 years or other types eligible for inclusion in the opinion of the investigator);
8. Known unstable mass or active radiographic evidence and symptoms of herniation severely limiting the recovery potential of the patient in the opinion of the investigator;
9. Known ruptured cerebral aneurysm, arteriovenous malformation, or vascular anomaly; hemorrhage from cerebral infarction, cerebral venous sinus embolization;
10. Has a platelet count < 100×109/L，(INR) > 1.5 or irreversible coagulopathy either due to medical condition or detected before screening;
11. Is taking new oral anticoagulants (such as dabigatran etexilate, rivaroxaban, apixaban, etc.) or low molecular weight heparin at the time of ICH onset;
12. In the opinion of the investigator is unstable and would benefit from supportive care rather than supportive care plus CN-105;
13. In the opinion of the investigator has any contraindication to the planned study assessments, including CT and MRI;
14. Severe renal insufficiency: creatinine clearance <30 mL/ min (Cockcroft-Gault formula), urea nitrogen and/or serum creatinine >1.5×ULN;
15. Is scheduled for surgical intervention throughout the trial period dose, including but not limited to hematoma evacuation (including minimally invasive and routine surgery), decompressive craniectomy, hematoma aspiration；
16. Clinically significant history of cardiovascular disease, including; (1) congestive heart failure (NYHA Class > 2); (2) unstable angina; (3) myocardial infarction in the past 12 months; (4) any need for treatment or interventional supraventricular arrhythmia or ventricular arrhythmia;
17. Has electrocardiogram (ECG) examination abnormalities deemed clinically significant by the investigator: for example, QTc interval prolongation during screening (male > 450 ms, female > 470 ms) (Note: QTc interval must be calculated according to Fridericia's criteria);
18. Subjects were disabled before disease onset (mRS ≥ 2)
19. Patients with past intracranial hemorrhage such as cerebral hemorrhage, subarachnoid hemorrhage, or cerebral infarction/transient ischemic attack (TIA, but excluding lucunar infarction);
20. Patients have other serious/severe acute or chronic mental illnesses, including recent (within the past 1 year) or current suicidal ideations or behaviors;
21. May increase the risks associated with participating in research or study drug management, or may interfere with the results of the study, or may interfere with the investigator's interpretation of laboratory abnormalities;
22. Patients are employees of the research center or family members directly related to the participants of this study, or subordinates who are not directly related to the trial but are subordinates of the trial, or are employed by the sponsor directly related to the trial;
23. Is predisposed to allergy or known allergy to any ingredient in the study drug;
24. Patients who have participated in other clinical trials or are participating in another interventional clinical study within 3 months prior to enrollment;
25. For other reasons, the investigator considered the subjects are inappropriate to be enrolled in the trial.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
AEs | 90±7 days
  Number and severity of AEs throughout the duration of the study;
SAEs | 90±7 days
  Number and severity of SAEs throughout the duration of the study;
Treatment-related mortality; | 90±7 days
  Treatment-related mortality throughout the duration of the study;
Deaths | Day14, Day30,Day90
  Rate of mortality at 14-day, 30-day, and 90-day ;
Incidence of cerebritis, meningitis, ventriculitis; | 90±7 days
  Incidence of cerebritis, meningitis, ventriculitis throughout the duration of the study;
Incidence of systemic infection associated with intracerebral hemorrhage | 90±7 days
  Incidence of systemic infection associated with intracerebral hemorrhage throughout the duration of the study;
The incidence of hematoma extension | 24-48 hour （Day2~Day3）
  The incidence of hematoma extension in 24-48 h after the first dose of study drug administration relative to baseline；

SECONDARY OUTCOMES:
Modified Rankin Scale(mRS) | Day90
  The proportion of patients alive and independent (mRS 0-2) on D90;
National Institutes of Health Stroke Scale (NIHSS) | 90±7 days
  During dosing neurological deterioration, defined as an increase of National Institutes of National Institutes of Health Stroke Scale (NIHSS) > 2 from baseline( unrelated to sedation)；
contrast head CT to evaluate progression of perihematomal edema; | screening, 24hour (Day2), 48hour (Day3) and 120hour (Day6),Day14
  At screening, 24h (D2), 48h (D3) and 120h (D6) after the first dose and D14, non-contrast head CT to evaluate progression of perihematomal edema;
Modified Rankin Scale(mRS) | Day30
  At D30 The proportion of patients alive and independent (mRS 0-2) and the distribution of mRS scores（shift analysis）at D30, D90;
Glasgow Coma Scale (GCS) | Day3, Day14
  Glasgow Coma Scale (GCS) assessment at D3, D14;
Barthel Index assessment | Day14, Day30, Day90
  Barthel Index assessment at D14, D30, D90;
Montreal Cognitive Assessment (MoCA) | Day2, Day30
  Montreal Cognitive Assessment (MoCA) Score at D2, D30;
MRI to evaluate the severity of neuronal injury and determine the progression of perihematomal edema respectively ； | screening, 48hour (Day3), 120hour (Day6)
  At screening, 48h (D3), 120h (D6) after the first dose of study drug, MRI to evaluate the severity of neuronal injury and determine the progression of perihematomal edema respectively ；

OTHER OUTCOMES:
Biomarker Outcome Measures: | screening, 48 hour(Day3), and 120 hour(Day6)
  Biomarker analysis at screening, 48 h(D3), and 120 h(D6) after the first dose:Cytokines and chemokines: G-CSF, GM-CSF, IFN-γ, IL-1α, IL-1β, IL-1ra, IL-6, IL-17A, IP-10/CXCL10, MCP-1/CCL2, MIP-1α/CCL3, TNF-α, VEGF-A; Molecular markers associated with the nervous system: ApoE, GFAP;
Genetic marker | screening
  Genotyping at screening:1ApoE gene polymorphism analysis;2SNP analysis of TOMM40-APOE locus

CONTACTS AND LOCATIONS:
Overall Officials: shuya Li, Study Director, Study Director — IRB of Beijing Tiantan Hospital,Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Beijing, China